CLINICAL TRIAL: NCT04929665
Title: Comparison of Ultrasound-guided Thoracic Paravertebral and Erector Spinae Plane Block Alone and in Combination on Analgesia After Video-assisted Thoracoscopic Surgery
Brief Title: Thoracic Paravertebral Block, Erector Spinae Plane Block, and in Combined Paravertebral-erector Spinae Block
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Atatürk Chest Diseases and Chest Surgery Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Musa Zengin, Principal investigator, Atatürk Chest Diseases and Chest Surgery Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: E.Kurul-E1-21-1688
Record Dates: First submitted 2021-06-10; First posted 2021-06-18 (Actual); Last update posted 2021-07-15 (Actual); Status verified 2021-07

CONDITIONS: Pain, Postoperative; Thoracic Surgery, Video-Assisted; Thoracic Paravertebral Block; Erector Spinae Plane Block
Keywords: Erector spinae block, Thoracic paravertebral block, VATS
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Thoracic Paravertebral Block (Active Comparator): In patients who are planned to have a thoracic paravertebral block, the needle will be advanced to the paravertebral area with ultrasound-guided in-plane technique. 20 ml of 0.25% bupivacaine will be injected into this area.
  Interventions: Procedure: Two different block and combination of these two blocks
- Erector spinae block (Active Comparator): Patients who are planned to have an erector spina block will be advanced to the interfacial area under the erector spinae muscle by ultrasound-guided in-plane technique. 20 ml of 0.25% bupivacaine will be injected into this area.
  Interventions: Procedure: Two different block and combination of these two blocks
- Thoracic Paravertebral block and Erector spinae Block (Active Comparator): In patients who are planned to have combined erector spinae block and thoracic paravertebral block, the needle will be advanced to the paravertebral area with ultrasound-guided in-plane technique. 10 ml of 0.25% bupivacaine will be given to this area. Then, with the same needle, return 1-2 cm from the paravertebral area and inject 10 ml of 0.25% bupivacaine into the interfacial area under the erector spinae muscle.
  Interventions: Procedure: Two different block and combination of these two blocks

INTERVENTIONS:
Procedure: Two different block and combination of these two blocks — Thoracic paravertebral block, erector spina block, and a combination of paravertebral block and erector spinae block will be applied to the patients under real-time ultrasound guidance.

SUMMARY:
Video-assisted thoracic surgery (VATS) has become a common procedure in thoracic surgery. Severe postoperative pain may be encountered in patients undergoing VATS. Analgesic methods such as thoracic paravertebral block (TPVB), intercostal block and erector spina plane block (ESPB) are widely used for VATS. Among these methods, ultrasound (US) guided TPVB is the most preferred method. Generally, comparisons are made between ESPB and TPVB in studies and the analgesic effect is evaluated. However, no research could be found in the literature combining ESPB and TPVB. The mechanisms of regional analgesia techniques used after thoracic surgery operations are also different from each other. Therefore, it may be possible to obtain a more effective analgesic effect in patients by combining the mechanism of action of TPVB and ESPB, as in the multimodal analgesia method. This study seeks to evaluate the effect of TPVB, ESPB and combined TPVB-ESPB pain after VATS.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 80 years old
* ASA physical status I-II-III
* BMI 18 to 30 kg/m2
* Elective video assisted thoracoscopic surgery

Exclusion Criteria:

* Patient refusing the procedure
* Emergency surgery
* Chronic opioid or analgesic use

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2021-07-01 (Actual); Study Completion 2021-07-13 (Actual)

PRIMARY OUTCOMES:
Pain scores [ Time Frame: 24 hours after the surgery] | 24 hours
  Pain will be assessed at rest and on coughing using the visual analog scale on a scale from 0 (no pain) to 10 (worst pain). Pain assessment will be done at 1st, 2nd, 4th, 8th, 16th and 24th hours after surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Musa Zengin, MD, Principal Investigator — Atatürk Chest Diseases and Chest Surgery Training and Research Hospital
Locations (1):
- Ankara Atatürk Chest Disease and Chest Surgery Training and Research Hospital, Keçiören, Ankara, Turkey (Türkiye)